CLINICAL TRIAL: NCT02608346
Title: Circulating Tumor DNA and Follow-up of BRCA1 Mutation Carriers (CirCa 01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2014-05
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Women With BRCA1 Germline Deleterious Mutation
Keywords: Circulating tumor DNA; BRCA1 mutation; Circulating tumor cells
MeSH Terms: conditions — Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood sampling (Other)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Patients will have a blood draw at each visit to the hospital,
  * with a maximum of 1 blood draw every 3 months, in absence of any abnormal clinical/radiological exam
  * with a maximum of 1 blood draw every week, in case of abnormal clinical/radiological exam that requires further investigation

SUMMARY:
BRCA1 carriers who are at high risk of developing either a relapse and/or a new cancer growth will be included. These patients will be followed up during 30 months (2,5 years) with mutated TP53 mutation detection or during 42 months (3,5 years) with mutated TP53 mutation detection and circulating tumor cells detection (CTC) performed at each hospital visit (for technical reason only patients included at Institut Curie will be proposed to participate to the CTC substudy).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with no evidence of any invasive tumor mass at inclusion (clinical and, if any, radiological exams)
2. Carriers of known germline BRCA1 deleterious mutation (a personal history of cancer is NOT mandatory).
3. Age ≥ 30 years for patient with personal previous history of cancer
4. Age ≥ 40 years for patient without personal previous history of cancer
5. Patient who a follow-up visit is scheduled in the including center at least once a year
6. Patient having health care insurance
7. Signed informed consent by patient

Exclusion Criteria:

1. Patient presenting with invasive tumor masses (e.g. stage IV cancer or localized cancer not yet surgically removed)
2. Carriers of germline BRCA1 variant of unknown significance
3. Carriers of germline BRCA2 deleterious mutation or variant
4. Individuals with a low risk of BRCA1-related tumor growth, i.e. women who underwent prophylactic bilateral mastectomy AND adnexectomy.
5. Any medical or other condition that in the Investigator's opinion rendered the patient unsuitable for this study
6. Patient deprived from ability to decide on her own.
7. Patient unable to have a regular follow up for geographical, social or psychological reasons.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity of plasma TP53 mutation detection as a test to detect any tumor growth (relapse and/or new tumor) during the follow-up of women known to carry BRCA1 germline mutation | Up to 42 months
  Sensitivity = % of patients with detectable levels of mutated TP53 ctDNA among those who experience a new tumor growth (relapse and/or new tumor).
Specificity of plasma TP53 mutation detection as a test to detect any tumor growth (relapse and/or new tumor) during the follow-up of women known to carry BRCA1 germline mutation | Up to 42 months
  Specificity = % of patients with undetectable levels of mutated TP53 ctDNA among those who don't experience a new tumor growth (diagnosed within 6 months after the blood draw).

SECONDARY OUTCOMES:
Positive predictive value for mutated TP53 ctDNA | Up to 42 months
  Positive predictive value = Probability of having a tumor growth (relapse and/or new tumor) when mutated TP53 ctDNA is detectable.
Negative predictive value for mutated TP53 ctDNA | Up to 42 months
  Negative predictive value = Probability of being without tumor growth when mutated TP53 ctDNA is not detectable.
Sensitivity of circulating tumor cells detection as a test to detect any tumor growth (relapse and/or new tumor) during the follow-up of women known to carry BRCA1 germline mutation | Up to 42 months
  Sensitivity = % of patients with detectable levels of circulating tumor cells among those who experience a new tumor growth (relapse and/or new tumor).
Specificity of circulating tumor cells detection as a test to detect any tumor growth (relapse and/or new tumor) during the follow-up of women known to carry BRCA1 germline mutation | Up to 42 months
  Specificity = % of patients with undetectable levels of circulating tumor cells among those who don't experience a new tumor growth (diagnosed within 6 months after the blood draw).
Positive predictive value for circulating tumor cells | Up to 42 months
  Positive predictive value = Probability of having a tumor growth (relapse and/or new tumor) when circulating tumor cells is detectable.
Negative predictive value for circulating tumor cells | Up to 42 months
  Negative predictive value = Probability of being without tumor growth when circulating tumor cells is not detectable.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves PIERGA, DR, Principal Investigator — Institut Curie
Locations (4):
- France (4):
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Hôpital René Huguenin - Institut Curie, Saint-Cloud
  - Institut Gustave ROUSSY, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).